CLINICAL TRIAL: NCT02523937
Title: Evaluation of Performances of Soluble Fibrin Assay in Exclusion of Pulmonary Embolism and Deep Venous Thrombosis
Brief Title: Evaluation of Soluble Fibrin in Thrombosis Exclusion
Acronym: FSET
Status: Completed | Type: Observational
Sponsor: Diagnostica Stago R&D (Industry)
Collaborators: Hôpital Louis Mourier (Other); Hopital Lariboisière (Other)
Responsible Party: Sponsor
Other Study IDs: FSET 2014-A00588-39
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Pulmonary Embolism (PE); Deep Vein Thrombosis (DVT)
Keywords: Pulmonary Embolism; Deep Venous Thrombosis; Soluble Fibrin; D-Dimers; Low and intermediate clinical probability
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — thrombus precursor protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen heparinized and citrated Poor Platelets Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group without PE or DVT: PE or DVT have to be confirmed or discarded by combining Wells score clinical probability, D-Dimer, and imaging tests.
  The criteria for exclusion of PE or DVT are:
  * low or intermediate clinical probability and D-dimer <0,50 µg/mL
  * low and moderate clinical probability and negative spiral computed tomography CT and/or proximal lower limb venous compression ultrasonography (US)
  * high clinical probability and negative CT and US.
  Soluble Fibrin assay will be performed in comparison with D-dimer assays.
  Interventions: Other: Soluble Fibrin
- Group with PE or DVT: PE or DVT have to be confirmed or discarded by combining Wells score clinical probability, D-Dimer, and imaging tests.
  The criteria for confirmation of PE or DVT are:
  * PE on spiral computed tomography (CT)
  * proximal deep vein thrombosis on ultrasonography (US).
  Soluble Fibrin assay will be performed in comparison with D-dimer assays.
  Interventions: Other: Soluble Fibrin

INTERVENTIONS:
Other: Soluble Fibrin — Evaluating the diagnostic performances of the assay in terms of sensitivity, specificity, negative and positive predictive values; from calculation of the area under the curve in comparison with the D-dimers.

SUMMARY:
The purpose of the study is to evaluate the performances of Soluble Fibrin assay for exclusion of Pulmonary Embolism and Deep Venous Thrombosis. Secondary objectives are to determine the threshold value from the ROC curves, the possible interest in the positive diagnosis of Venous Thromboembolism (VTE), and to verify the absence of influence of age on the SF results.

DETAILED DESCRIPTION:
Rationale. Pulmonary embolism (PE) is a major public health problem. D-dimer (D-Di) assay is useful to exclude VTE (DVT and PE) but not specific, requiring irradiating and expensive imaging tests. Preliminary results suggest that the Soluble Fibrin (SF) assay has a sensitivity comparable to the D-Di one, but a higher specificity and thus would limit the use of imaging tests.

Main objective. To evaluate the performances of Soluble Fibrin assay in terms of sensitivity, specificity, negative and positive predictive values for exclusion of Pulmonary Embolism and Deep Venous Thrombosis, in comparison with the D-Dimer test. To determine the threshold value from the ROC curves.

Patients. Inclusion criteria: patients 18 years or older, referred to the Emergency or Internal Medicine Units, for clinically suspected of PE or DVT.

The study was conducted in compliance with French regulation after ethics approval, the authorization for processing personal data (Commission Nationale de l'Informatique et des Libertés, 8, rue Vivienne CS 30223 75083 Paris Cedex 02) decision DR-2015-174 was obtained in April 2015. A preliminary study was performed from April 2015 to September 2015 to define the exclusion criteria.

Comparison with the D-Dimer test. Plasma D-dimer (D-Di) and soluble fibrin are measured in case of low and intermediate clinical probability.

Patients will be classified in two groups, as having or not having PE or DVT on predefined criteria according to the recent guidelines of the European Society of Cardiology by physicians who will be unaware of the SF assay result. PE and DVT have to be confirmed or excluded by the reference algorithm combining clinical probability, D-Dimer, and imaging tests with three month-follow up. The patient who could not be contacted after three months are included in the study and taken into account with the mention "without follow up".

SF Assays. Soluble fibrin is measured by one site, using prototype assays, on both citrated and heparinized frozen plasma taken at baseline. Staff in charge of the assays are not aware of the clinical and diagnosis decisions.

Statistical Analysis of results. The results of D-dimer and Soluble Fibrin assays for the exclusion of PE and DVT will be interpreted on the basis of sensitivity, specificity, negative and predictive values. The ROC curve will be built, the area under the curve will be calculated with its confidence interval. The most suitable threshold will be determined from the curve. Then the diagnosis performances of SF assay will be calculated according to the usual calculations.

The patients under anticoagulant treatment or with an activation of coagulation from known cause are included in the study but analyzed separately.

Number of participants required. A statistical analysis was realized before starting the study. The inclusion of 50 patients with a positive diagnostic of PE or DVT and about 350 patients with an exclusion of PE or DVT will allow calculation of the diagnosis performances of the SF assay and of the area under the ROC curve with an accuracy of 5%. Duration of the study. The total duration of the study is 12 months and up to 18 months if the number of patients could not be obtained.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-opposition to participate in the evaluation,
* outpatients from Emergency or Internal Medicine Units,
* clinically suspected of PE or DVT.

Exclusion Criteria:

* patients under 18 years old,
* patients with opposition to participate in the evaluation,
* patients with contraindication to iodinated contrast media.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients from Emergency or Internal Medicine Units, in a French Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 863 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Performances of the Soluble Fibrin Assay for the exclusion of PE and DVT | 24 Months
  Determination of the sensitivity and specificity of the Soluble Fibrin Assay to calculate the area under the ROC curve for exclusion of PE and DVT. The most suitable threshold will be determined from the curve.

SECONDARY OUTCOMES:
Threshold of the Soluble Fibrin assays for the exclusion of PE and DVT | 24 Months
  The most suitable threshold will be determined from the curve. Then the exclusion performances of SF assays will be calculated according to the usual calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mahe, MD, PhD, Principal Investigator — Université of Paris 7 - Paris Diderot; Geneviève Contant, PhD, Study Director — Diagnostica Stago
Locations (1):
- Internal Medecine Unit - Adults Pole and Hematology Laboratory Hôpital Louis Mourier (AP-HP), Colombes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirshahi S, Soria C, Kouchakji B, Kierzek G, Borg JY, Varin R, Chidiac J, Drouet L, Mirshahi M, Soria J. New combinational assay using soluble fibrin and d-dimer determinations: a promising strategy for identifying patients with suspected venous thromboembolism. PLoS One. 2014 Mar 24;9(3):e92379. doi: 10.1371/journal.pone.0092379. eCollection 2014. PMID 24664182